CLINICAL TRIAL: NCT01513616
Title: Mechanisms of Dyspnea Relief Following Exercise Training in COPD
Brief Title: The Impact of Pulmonary Rehabilitation on Dyspnea in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMED-986-06
Record Dates: First submitted 2012-01-11; First posted 2012-01-20 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; dyspnea; exercise; measurement; respiratory physiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary rehabilitation (Experimental): A supervised 8-wk outpatient pulmonary rehabilitation program consisting of multi-modality exercise training and COPD self-management education.
  Interventions: Other: Pulmonary rehabilitation
- Usual care control (Sham Comparator): An 8-wk control period consisting of usual medical care which included optimization of respiratory medications, instructions on how best to manage COPD, standard access to treatment in the event of an exacerbation, self-management education.
  Interventions: Other: Pulmonary rehabilitation; Other: Usual care

INTERVENTIONS:
Other: Pulmonary rehabilitation — 8-week program, 3 supervised session per week
Other: Usual care — An 8-week control period (includes optimization of respiratory medications, instructions on how best to manage COPD, standard access to treatment in the event of an exacerbation, self-management education)
  Arms: Usual care control

SUMMARY:
Dyspnea (respiratory discomfort) and activity limitation are the most common symptoms of chronic obstructive pulmonary disease (COPD) and contribute importantly to a perceived poor quality of life. Recent international guidelines have stressed the importance of dyspnea alleviation and improvement exercise tolerance as a means of enhancing quality of life and other long term outcomes in this population. Modern pharmacotherapy is the first step in symptom management but the overall impact of bronchodilator therapy is relatively small. Exercise training remains the most effective treatment for ameliorating dyspnea and improving exercise endurance and was the main focus of this study.

The main objectives of the study were:

1. To conduct and compare detailed studies of respiratory mechanics during cycle exercise before and after exercise training (EXT) compared with an untrained control group. By multiple regression analysis, the investigators will establish the main contributors to dyspnea relief after EXT.
2. To compare the magnitude of change in endurance during constant work rate cycle exercise with those measured during walk tests and the endurance shuttle walk test after EXT relative to control. To evaluate which test (constant work rate cycle, six-minute walk test, or endurance shuttle walk test) is the most sensitive test for measuring changes in endurance after EXT versus control.
3. To compare the change in standardized dyspnea ratings (Borg Scale) during constant-load cycling with a variety of other activity-related dyspnea questionnaires. To evaluate which of these measurements is the most sensitive for examining changes in perceived discomfort during exercise.
4. To evaluate the contribution of psychological factors (anxiety, fear, respiratory panic, self-efficacy) to the perceived improvement of symptoms following EXT. The investigators will use multiple regression analysis to examine associations between changes in perceived dyspnea and changes in anxiety and self-efficacy measured by validated questionnaires and Borg intensity ratings?

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD
* clinically stable
* presence of activity-related dyspnea (Baseline Dyspnea Index < 9)
* 40-80 years of age

Exclusion Criteria:

* other significant disorders or diseases that could interfere with conduct of the intervention or tests
* body mass index < 18 or > 40 kg/m2

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Exertional dyspnea intensity | 8 weeks
  Post-intervention comparisons (pulmonary rehabilitation vs. usual care control) of dyspnea measurements (i.e., Borg ratings at a standardized time during high-intensity constant-work rate cycle exercise testing)

SECONDARY OUTCOMES:
Multidimensional measurements of dyspnea and physiological measurements | 8 weeks
  Activity-related dyspnea: MRC dyspnea scale, Transition Dyspnea Index, CRQ dyspnea component, SGRQ activity component
Dyspnea-related anxiety | 8 weeks
  Intensity of dyspnea-related anxiety measured during cycle exercise testing (Borg scale)
disease-specific self-efficacy | 8 weeks
  COPD Self-Efficacy Score
Pulmonary function | 8 weeks
  Detailed measurements of pulmonary function: spirometry, body plethysmography, diffusing capacity, maximal respiratory pressures
Cardiopulmonary exercise test measurements | 8 weeks
  Physiological measurements obtained during cycle exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit at Kingston General Hospital, Kingston, Ontario, Canada